CLINICAL TRIAL: NCT04612543
Title: Randomized, Controlled Clinical Evaluation of Extensive Direct Composite Restorations With Polyethylene Fiber in the First Permanent Molars of Children
Brief Title: Clinical Evaluation of Extensive Direct Composite Restorations With Polyethylene Fiber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Semanur Özüdoğru, Assistant Professor, Kafkas University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KafkasU
Record Dates: First submitted 2020-10-26; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Dental Caries Extending Into Dentin
Keywords: Composite resin; Clinical Evaluation; Polyethylene Fiber; First Permanent Molars; Extensive carious

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genial Posterior Composite with Polyethylene fiber (Active Comparator): The enamel and dentin were conditioned with bonding procedure.After bonding procedures, remaining tooth composite resin walls were created and cured for 20 s. Prepared ribbond fiber pieces, 2-mm-wide approximately 12mm-long, (Ribbond Thinner, Higher, Modulus - Ribbond Inc,Seattle) were wetted with an unfilled resin for 2 minutes at a non-light environment. The inner surfaces of the prepared class I cavity were lined with flowable resin. After removing the excess resin, pre-wetted polyethylene fiber was condensed circumferentially and embedded with a hand instrument into the bed of unpolymerized flowable composite and then polymerized for 20 seconds with Light Emitting Diodes. After curing for 20 s, composite resin was applied to the rest of the cavity incrementally, each increment was cured for 20 seconds. Finally, the restoration was shaped with finishing diamonds and silicon instruments.
  Interventions: Device: Genial Posterior Composite with Polyethylene Fiber; Device: Genial Posterior Composite
- Genial Posterior Composite (Active Comparator): The enamel and dentin were conditioned with bonding procedure using an applicator, left undisturbed for five to 10 seconds, and then dried thoroughly for five seconds with oil-free air under air pressure, Genial Direct Posterior resin was applied with the incremental technique (2 mm thick layers) and light-cured for 20 seconds. Finally, the restoration was shaped with finishing diamonds and silicon instruments
  Interventions: Device: Genial Posterior Composite with Polyethylene Fiber; Device: Genial Posterior Composite

INTERVENTIONS:
Device: Genial Posterior Composite with Polyethylene Fiber — Placing restorations,Genial Posterior Composite with Polyethylene Fiber, after bonding procedures, remaining tooth composite resin walls were created and cured for 20 s. Prepared ribbond fiber pieces, 2-mm-wide approximately 12mm-long, (Ribbond Thinner, Higher, Modulus, Ribbond Inc,Seattle) were wetted with an unfilled resin for 2 minutes at a non-light environment. The inner surfaces of the prepared class I cavity were lined with flowable resin. After removing the excess resin, pre-wetted polyethylene fiber was condensed circumferentially and embedded with a hand instrument into the bed of unpolymerized flowable composite and then polymerized for 20 seconds with Light Emitting Diodes. After curing for 20 s, composite resin was applied to the rest of the cavity incrementally, each increment was cured for 20 seconds. Finally, the restoration was shaped with finishing diamonds and silicon instruments.
  Other Names: Micro hybrid composite with Polyethylene Fiber
Device: Genial Posterior Composite — Placing Genial Posterior Composite, the enamel and dentin were conditioned with bonding procedure using an applicator, left undisturbed for five to 10 seconds, and then dried thoroughly for five seconds with oil-free air under air pressure, Genial Direct Posterior resin was applied with the incremental technique (2 mm thick layers) and light-cured for 20 seconds. Finally, the restoration was shaped with finishing diamonds and silicon instruments
  Other Names: Micro hybrid composite

SUMMARY:
The aim of this clinical trial was to compare the clinical performances of composite resin restorations with/without the polyethylene fiber to the first permanent molar teeth with extensively carious pediatric patients. A total of 75 restorations with (FC; n=38)or without (C; n=37) fiber were placed in the first permanent molar teeth.

Restorations were evaluated at baseline-6-12-18 months according to the modified-USPHS criteria. Data were analyzed with Chi-Square and Cochran's Q (p<0.05).

DETAILED DESCRIPTION:
Fiber reinforced composite restorations developed in recent years have been presented to improve the negative properties of composite resin systems applied by the traditional method thanks to the fact that the fibers act as a crack stopper, reduce polymerization shrinkage by decreasing the the mass of composite resin material between the remaining dentin structure and the fiber. Many authors having conducted tremendous experience in this field of research have reported that the polyethylene fiber is an innovative approach because it not only increases the flexural strength but also improves fracture toughness. Its woven fiber orientation provides the stresses to be dispersed throughout the restoration, and therefore reinforces the restoration and the remaining tooth structure in multiple directions.

ELIGIBILITY:
Inclusion Criteria:

* no hypoplasia or any tissue abnormality in the teeth,
* deep dentin caries with three tubercle loss in the teeth, need of three surface restorations with coverage of at least two adjacent cusps.
* no evidence for pulpal complications
* in occlusion

Exclusion Criteria:

* partly erupted teeth;

  -.absence of adjacent and antagonist teeth
* poor periodontal status;
* adverse medical history;
* potential behavioral problems.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Marginal adaptation | From baseline to 18 months the change of restorations was evaluated
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria Observers evaluated the restorations was performed using the modified United State Public Health Service criteria which was evaluated by 2 independent clinicians. Visual inspection with a mirror at 18 inches was performed. A score means the higher score of clinical acceptability while C and D score means that the restoration has failed and needs to be replaced. Alpha 1: Harmonious outline Alpha 2: Marginal gap with discoloration (removable)
marginal discoloration | From baseline to 18 months the change of restorations was evaluated
  Alpha: No discoloration anywhere along the margin between the restoration and the adjacent tooth. Bravo: Slight discoloration along the margin between the restoration and the adjacent tooth. Charlie: The discoloration penetrated along the margin of the restorative material in a pulpal direction
retention rate | From baseline to 18 months the change of restorations was evaluated
  Alpha 1:Clinically excellent Alpha 2: Clinically good with slight deviations from ideal performance, correction possible without damage of tooth or restoration Bravo: Clinically sufficient with few defects, corrections or repair of the restoration possible Charlie: Restoration is partially missed Delta: Restoration is totally missed
anatomic form | From baseline to 18 months the change of restorations was evaluated
  Alpha 1: Continuous with existing anatomical form Alpha 2: Slightly discontinuous due to some chipping on the proximal ridge Bravo: Discontinuous with existing anatomical form due to material loss but proximal contact still present Charlie: Proximal contact is lost with ridge fracture.
color change | From baseline to 18 months the change of restorations was evaluated
  Alpha: The restoration matches the adjacent tooth structure in color and translucency.
  Bravo: Light mismatch in color, shade or translucency between the restoration and the adjacent tooth. Charlie: The mismatch in color and translucency is outside the acceptable range of tooth color and translucency
  Alpha: The restoration matches the adjacent tooth structure in color and translucency.
  Bravo: Light mismatch in color, shade or translucency between the restoration and the adjacent tooth. Charlie: The mismatch in color and translucency is outside the acceptable range of tooth color and translucency

CONTACTS AND LOCATIONS:
Overall Officials: SEMANUR ÖZÜDOĞRU, Ass.. Prof, Study Director — Kafkas University School of Dentistry
Locations (1):
- Kafkas University School of Dentistry, Kars, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Deliperi S, Alleman D, Rudo D. Stress-reduced Direct Composites for the Restoration of Structurally Compromised Teeth: Fiber Design According to the "Wallpapering" Technique. Oper Dent. 2017 May/Jun;42(3):233-243. doi: 10.2341/15-289-T. PMID 28467261
- [Background] Candan U, Eronat N, Oncag O. Clinical performance of fiber-reinforced nanofilled resin composite in extensively carious posterior teeth of children: 30-month evaluation. J Clin Pediatr Dent. 2013 Fall;38(1):1-6. doi: 10.17796/jcpd.38.1.q352786473372282. PMID 24579274
- [Background] Garoushi S, Lassila LV, Tezvergil A, Vallittu PK. Static and fatigue compression test for particulate filler composite resin with fiber-reinforced composite substructure. Dent Mater. 2007 Jan;23(1):17-23. doi: 10.1016/j.dental.2005.11.041. Epub 2006 Jan 18. PMID 16414110